CLINICAL TRIAL: NCT04801199
Title: Prospective, Randomized, Double Blind, Parallel Group, Two Arm, Comparative, Multicenter, Clinical Study to Compare Efficacy and Safety of Oral CPL-2009-0031 140 mg of Cadila Pharmaceutical Limited, India Against Innovator Sitagliptin 100 mg in Patients With Uncontrolled Type-2 Diabetes Mellitus (T2DM)
Brief Title: Effect of CPL-2009-0031 in the Treatment of Patients With Uncontrolled Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cadila Pharnmaceuticals (Industry)
Collaborators: New Millennium Indian Technology Leadership Initiative (NMITLI) program of Council of Scientific and Industrial Research, India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRSC18005
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Uncontrolled Type 2 Diabetes Mellitus
MeSH Terms: interventions — Sitagliptin Phosphate

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Double Blind, Parallel Group, Two arm, Comparative, Multicenter, controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigator, patient, study staff, data monitors and database personnel will be blinded to the study treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPL-2009-0031 140 mg (Experimental): Single dose, Oral tablet containing 140 mg of CPL-2009-0031, Once daily for 36-weeks
  Interventions: Drug: CPL-2009-0031 140 mg
- Sitagliptin 100 mg (Active Comparator): Single dose, Oral tablet containing 100 mg of Sitagliptin, Once daily for 36-weeks
  Interventions: Drug: Sitagliptin 100mg

INTERVENTIONS:
Drug: CPL-2009-0031 140 mg — Patients will receive OD CPL-2009-0031 140 mg for 36 weeks with or without breakfast with a glass of water.
  Arms: CPL-2009-0031 140 mg
Drug: Sitagliptin 100mg — Patients will receive OD Sitagliptin 100 mg for 36 weeks with or without breakfast with a glass of water.
  Arms: Sitagliptin 100 mg

SUMMARY:
This trial is a Phase-III, Prospective, Randomized, Double Blind, Parallel Group, Two arm, Comparative, Multicenter, controlled clinical trial to determine the efficacy, safety, and tolerability of oral CPL-2009-0031 140 mg in comparison with Sitagliptin 100 mg in patients with Uncontrolled Type-2 Diabetes Mellitus (T2DM).

DETAILED DESCRIPTION:
In this phase-III trial, after due consent and completing initial 2-weeks of placebo run-in period with diet, exercise and counseling, eligible patients with uncontrolled T2DM will be randomized in balance to receive either once daily oral CPL-2009-0031 140 mg or Sitagliptin 100 mg.

After completing 12 weeks of study post-randomization for regulatory submission, patients will be instructed for continuation of extension phase of treatment and follow up upto 36 weeks.

HbA1c will be measured at screening, baseline, 12 weeks, 24 weeks and 36 weeks of treatment. While, Fasting Blood Sugar (FBS) and Postprandial Blood Sugar (PPBS) measurement will be performed every 2 weeks.

The enrolled patients will be monitored for safety (AE and SAE) throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult patient of 18-65 years with uncontrolled type 2 diabetes Mellitus (T2DM).
* Patients with HbA1c ≥ 7 to 10 and those on oral hypoglycemic agents ≤ 2 other than Insulin and Gliptins.
* BMI in the range of 18.5 - 35 kg/m2.
* All patients must be willing to give informed consent and can understand & complying protocol requirement.
* Patients who are in good health at the time of entry into the study as determined by medical, medication and hypersensitivity histories, clinical examination, vital sign measurements, chest X-ray, 12-lead ECG measurement and clinical judgment of the investigator.
* Documented negative test for human immuno virus (HIV), Hepatitis B surface antigen (HBsAg) and Hepatitis C virus (HCV).

Exclusion Criteria:

* Those who are on insulin and not ready for wash out of 3 months.
* Those who are on gliptin and not ready for wash out of 3 months.
* Those with a history of severe ketosis, diabetic coma or pre-coma, or type 1 diabetes.
* Those scheduled for or who had undergone surgery.
* Those with a severe infection or serious injury
* Pregnant and lactating women.
* Hypersensitivity and contraindication to DPP-IV inhibitors or excipients of investigational drug formulation.
* Hypertensive patients with blood pressure ≥160/100 mm of Hg.
* History of ischemic heart disease (as evident from ECG), stroke and/or transient ischemic attack.
* Debilitating neurological or psychiatric disorders
* History or currently consuming abusing drugs or alcohol.
* Serious hepatic or renal impairment (liver dysfunction as evidenced by SGPT/SGOT level of 2.5 X ULN and renal dysfunction as evidenced by creatinine level 2.5 X ULN).
* Patient with abnormal clinical chemistry, hematology or urinalysis results that are considered clinically significant by the investigator or the sponsor.
* Patient has any concurrent illness which, in the opinion of the investigator or coinvestigator, may interfere with treatment or evaluation of safety or completion of this study.
* In the investigator's judgment, the patient is unable to adhere to the treatment regimen, protocol procedures or study requirements.
* Participation in another clinical trial in the past 3 months.
* Patients with history of smoking or currently having smoking habit will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2020-01-26 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c level | Baseline, 12 weeks, 24 weeks and 36 weeks from onset of therapy
  To evaluate HbA1c levels between oral CPL-2009-0031 140 mg and oral Sitagliptin 100 mg

SECONDARY OUTCOMES:
Fasting Blood Sugar (FBS) level | Every 2 week till 12 weeks and every 4 weeks between 12 weeks to 36 weeks from onset of therapy
  To compare Fasting Blood Sugar between oral CPL-2009-0031 140 mg and oral Sitagliptin 100 mg
Postprandial Blood Sugar (PPBS) level | Every 2 week till 12 weeks and every 4 weeks between 12 weeks to 36 weeks from onset of therapy
  To compare Fasting Blood Sugar between oral CPL-2009-0031 140 mg and oral Sitagliptin 100 mg
Frequency of Serious Adverse Events | From randomization to end of 12 week, 24 week and 36-weeks therapy
  Determination of safety and tolerability of CPL-2009-0031 140 mg versus Sitagliptin 100 mg based on Frequency of serious adverse events
Number of hypoglycemic events | From randomization to end of 12 week, 24 week and 36-weeks therapy
  Determine number and severity of hypoglycemic events of CPL-2009-0031 140 mg versus Sitagliptin 100 mg
Frequency of adverse events | From randomization to end of 12 week, 24 week and 36-weeks therapy
  Determine frequency and severity of adverse events of CPL-2009-0031 140 mg versus Sitagliptin 100 mg

CONTACTS AND LOCATIONS:
Overall Officials: Anil Avhad, MBBS, Study Director — Cadila Pharmaceutical Limited
Locations (12):
- India (12):
  - A C Subba Reddy Government Medical College and Hospital, Nellore, Andhra Pradesh
  - Downtown Hospital, Guwahati, Assam
  - SSG Hospital, Vadodara, Gujarat
  - Bangalore Diabetes Centre, Bangalore, Karnataka
  - Dhadiwal Hospital, Nashik, Maharashtra
  - Ashirwad Hospital & Research Centre, Ulhasnagar, Maharashtra
  - S.P. Medical College and A.G. Hospital, Bikaner, Rajasthan
  - Bhandari Clinic & Research Centre, Jaipur, Rajasthan
  - Sanjivini Lung Centre, Lucknow, Uttar Pradesh
  - Nilratan Sircar Medical College & Hospital, Kolkata, West Bengal
  - Life Line Diagnostic Centre cum Nursing Home, Kolkata, West Bengal
  - Apollo Hospital International Ltd, Gandhinagar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trial database uploaded on Clinical Trial Registry of India (CTRI) — http://www.ctri.nic.in/Clinicaltrials/pdf_generate.php?trialid=32963&EncHid=&modid=&compid=%27,%2732963det%27